CLINICAL TRIAL: NCT03222947
Title: Identification of New Genes Involved in the Taybi-Linder Syndrome.
Brief Title: New Variants Involved in Taybi-Linder Syndrome
Acronym: NewViTALS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0774
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Taybi Linder Syndrome; Genetic Syndrome
MeSH Terms: conditions — Microcephalic osteodysplastic primordial dwarfism, type 1; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Deoxyribonucleic acid of patients obtained either from blood samples (lymphocytes) or foetal tissue sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Taybi-Linder index cases: Taybi-Linder index cases who have already consented for the (re)use of their DNA samples for medical research.
  Interventions: Genetic: Deoxyribonucleic acid analysis
- Blood relatives of Taybi-Linder index cases: Blood relatives of Taybi-Linder index cases who have already consented for the (re)use of their DNA samples for medical research.
  Interventions: Genetic: Deoxyribonucleic acid analysis

INTERVENTIONS:
Genetic: Deoxyribonucleic acid analysis — This study consists in the high throughput exome sequencing and subsequent genetic bio-analysis of 19 deoxyribonucleic acid samples from 6 families, already collected and consented, including patients diagnosed with a Taybi-Linder syndrome and their relatives (parents and/or siblings).

SUMMARY:
Taybi-Linder syndrome (TALS, OMIM 210710) is a rare autosomal recessive disorder belonging to the group of microcephalic osteodysplastic primordial dwarfisms (MOPD). This syndrome is characterized by short stature, skeletal anomalies, severe microcephaly with brain malformations and facial dysmorphism, and is caused by mutations in RNU4ATAC. Although RNU4ATAC-associated TALS is a recognizable phenotype, an atypical presentation is sometimes observed, thus expanding the clinical spectrum (TALS-like phenotype).

This study aims to identify new variants involved in Taybi-Linder syndrome and associated phenotypes (i.e.TALS-like).

This non interventional study will be performed on patients with no proven mutation of RNU4ATAC and their blood relatives (19 samples total) by high throughput sequencing and genetic analysis of already collected deoxyribonucleic acid samples.

Altogether, such a study will allow a better understanding of the molecular mechanisms responsible for the Taybi-Linder syndrome and Taybi-Linder syndrome-like phenotypes as well as the pathophysiology of these devastating forms of microcephalic dwarfism.

ELIGIBILITY:
Inclusion Criteria:

* foetus or young children diagnosed with a Taybi-Linder or Taybi-Linder like syndrome, with no RNU4ATAC mutation (index case)
* aged 20 weeks pregnant to 18 years old
* parents or sibling of the index cases, with informed consent for the analysis of both their DNA sample and the one of the index case.

Exclusion Criteria:

* no informed consent for the use of genetic samples for medical research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with a Taybi-Linder or Taybi-Linder like syndrome and their blood relatives.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Identification of new variants involved in the Taybi-Linder syndrome | Collection at time of diagnosis = less than one day
  A genetic high throughput exome capture sequencing of 19 deoxyribonucleic acid samples from patients diagnosed with a Taybi-Linder like syndrome and their blood relatives

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Génétique Clinique, Groupement Hospitalier Est, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No